CLINICAL TRIAL: NCT05024474
Title: Effects of Inspiratory Muscle Training After Covid-19
Brief Title: Effects of Inspiratory Muscle Training After Covid-19 (ReCOV)
Acronym: IMT-ReCov
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Nygren-Bonnier, Physiotherapist, Senior lecturer and Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMT-ReCOV
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Covid-19; Respiratory Complication; Post-Acute Covid-19 Syndrome
Keywords: Inspiratory muscle training; Physiotherapy; Rehabilitation; Maximal inspiratory pressure; Respiratory Muscle Training
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The interventions were not possible to mask for participants or health care professionals (physiotherapist leading interventions). The physiotherapists who performed the tests after interventions were blinded to the group allocation. All data were coded and group assignment was blinded for the outcome analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: inspiratory muscle training + physical exercise (Experimental): Inspiratory muscle training (IMT) twice a day for 8 weeks combined with a physical exercise program at least two times a week for 8 weeks.
  Interventions: Other: Inspiratory muscle training (IMT); Other: Physical exercise
- Active control: physical exercise (Active Comparator): A physical exercise program at least two times a week for 8 weeks.
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Inspiratory muscle training (IMT) — Inspiratory muscle training (IMT) at 20-50 % of maximal inspiratory pressure (MIP), 2 x 30 repetitions, twice a day for 8 weeks.
  Arms: Intervention: inspiratory muscle training + physical exercise
Other: Physical exercise — A physical exercise program at least two times a week for 8 weeks. Including strength, aerobic and mobility exercises.

SUMMARY:
Initially, it was suspected that Covid-19 would primarily affect the airways, but several studies have now shown that it is a disease with multisystem manifestations. Covid-19 has the potential to affect physical, cognitive, and psychological functions in multiple ways. It has been clear that a significant proportion of patients with Covid-19 develop long-term symptoms. The term post-acute Covid-19 syndrome (PACS) is now used to describe the wide range of prolonged symptoms following the infection. Patients who have been in hospital for Covid-19 for a long time may need specialized rehabilitation, however, also non-hospitalized patients with mild symptoms may need specific rehabilitation to be able to meet the complex symptoms and problems that may arise. Previous studies on the recovery and rehabilitation after other coronavirus shows the importance to develop tailored interventions so that these patients receive appropriate rehabilitation

The aim of this study is to evaluate the effects of inspiratory muscle training on adult patients with PACS and decreased respiratory muscle strength.

A randomized controlled trial will be used. A total of 90 adult patients with PACS and 80 % or less of predicted value in inspiratory muscle strength (maximal inspiratory pressure) will be eligible for enrollment. Patients will be randomized either to an intervention group or a control group. The intervention will consist of inspiratory muscle training performed twice daily for 8 weeks. This will be combined with an 8-week physical exercise training program. The control group will perform the same physical exercise training according to standard care. All measurements will be performed at baseline and after 8 weeks.

Primary outcome is maximal inspiratory pressure. Secondary outcomes are: Maximal expiratory pressure, pulmonary function, physical capacity, physical activity, respiratory status and symptoms, health-related quality of life, work ability, fatigue, self-reported outcome measure of physical function and voice function.

Covid-19 has the potential to affect physical, cognitive, and psychological functions in multiple ways and lead to a negative impact on quality of life in the long-term perspective. Therefore, development of a rehabilitation program with specific tailored interventions will be necessary to improve physical and psychological function, as well as health-related quality of life and work ability.

DETAILED DESCRIPTION:
Introduction:

Covid-19 was declared a global pandemic in March 2020 by the World Health Organization (WHO). So far (August 2021), there are over 1 100 000 confirmed cases and over 14 000 deaths in Sweden. Initially, it was suspected that Covid-19 would primarily affect the airways, but several studies have now shown that it is a disease with multisystem manifestations. The impact of the virus ranges from an asymptomatic infection to a severe and life-threatening disease that can affect the cardiac, renal gastrointestinal, nervous, endocrine, and musculoskeletal systems. Therefore, Covid-19 has the potential to affect physical, cognitive, and psychological functions in multiple ways. It has been clear that a significant proportion of patients with Covid-19 develop long-term symptoms. Signs and symptoms may arise from any system in the body, often with significant overlap, and may develop over time. The term post- acute Covid-19 syndrome (PACS) is now used to describe the wide range of prolonged symptoms following the infection.

Fatigue, decreased physical and psychological function have been reported in the initial recovery phase, but still little is known on the long-term consequences. Patients who have been in hospital for Covid-19 for a long time may need specialized rehabilitation, however, also non-hospitalized patients with mild symptoms may need specific rehabilitation to be able to meet the complex symptoms and problems that may arise. Previous studies on the recovery and rehabilitation after other coronavirus shows the importance to develop tailored interventions so that these patients receive appropriate rehabilitation with a multi-professional approach throughout the whole care chain. Some studies suggest that the rehabilitation should be similar to pulmonary rehabilitation, but since a lot of patients often have symptoms from different organ systems this is not yet fully investigated and needs to be addressed from different perspectives. A study by Liu et al (2020), showed that 6 weeks of physical exercise and respiratory muscle training improved lung function and physical capacity compared to a control group in elderly patients after Covid-19.

At the Karolinska University Hospital there is a specialized multidisciplinary and multi-professional approach aiming to follow up patients who have been hospitalized. However, from mid-2020 and onwards, referrals from primary care have significantly increased. This includes patients who have never been hospitalized but with varying symptoms from several organs that have lasted for more than 3 months.

This study is part of a bigger research project (ReCoV) and is integrated with the clinical follow-up and linked research project of patients who have been hospitalized or referred from primary care

Hypothesis: The overall hypothesis of the hole research project is that physical and physiological function, work ability and HRQoL are important factors for recovery after Covid-19 which can be improved by individual tailored rehabilitation.

The aim of this study is to evaluate the effects of inspiratory muscle training (IMT) on physical and psychological function, work ability and HRQoL in patients with decreased respiratory muscle strength after Covid-19.

Methods:

To evaluate the effects of IMT, a randomized controlled trial design will be used.

Participants:

Patients with PACS above 18 years old (N=90) with 80% or less of predicted value in maximal inspiratory pressure (MIP) are eligible for participation in the study.

Procedure:

Baseline assessment before the intervention period will be performed at an outpatient visit at Karolinska university hospital. After baseline assessment participants will be randomized to either an intervention group or to an active control group using random permuted blocks. The intervention will take place at the physiotherapy outpatient clinic at the hospital or at a primary care facility and in the participants' homes. The intervention group will perform IMT twice daily (two sets of 30 receptions) at home during 8 weeks with a resistance of 20-50 % of MIP using an inspiratory muscle trainer (Threshold or digital advice). Follow-up of execution and increase in intensity during IMT will be conducted weekly by the physiotherapist. This will be combined with an 8-week physical exercise program including aerobic, strength and mobility exercises which will be performed at the care facility and at home at least two times a week. The active control group will perform the same physical exercise program according to standard care.

Outcome assessment:

All measurements will be performed at baseline and after the intervention period (8 weeks).

Primary outcome is maximal inspiratory pressure (MIP) and secondary outcomes are: maximal expiratory pressure (MEP), lung function, physical capacity (6-min walk test), Chair stand test, physical activity, respiratory status and symptoms, health-related quality of life, work ability, fatigue, self-reported outcome measure of physical function and voice function.

Statistical analyses:

Descriptive statistics will be presented as mean (standard deviation), median (interquartile range), and proportions, as appropriate. Depending on the level and distribution of the data, parametric or non-parametric methods will be applied to.

Originally, longitudinal group differences were to be analyzed using linear mixed models. A sample size calculation indicated that 36 participants per group would be required to detect a 10% difference in maximal inspiratory pressure (MIP), with an additional 25% added to account for potential dropouts, resulting in a target of 45 participants per group.

However, due to a lower-than-expected number of included participants and unmet assumptions for linear mixed models, the analysis plan has been revised. The updated plan includes an intention-to-treat analysis to assess between-group differences in outcome variables. Depending on the type of outcome variable, multiple linear or logistic regression models will be used, with the outcome variable as the dependent variable. Missing post-intervention data will be imputed using multiple imputation via the "mice" package in R.

Clinical significance:

Covid-19 has the potential to affect physical, cognitive, and psychological functions in multiple ways and lead to a negative impact on quality of life in the long-term perspective. Therefore, development of a rehabilitation program with specific tailored interventions will be necessary to improve physical and psychological function, as well as health-related quality of life and work ability.

Covid-19 is a new disease and large knowledge gaps need to be filled. Previous studies indicate that the patients are affected at several levels and a rehabilitation period is necessary. It is of great importance that data is collected systematically and standardized. If significant effects occur, the possibility to generalize the results to other individuals with Covid-19, are promising. The physical interventions may thus improve the ability to adjust to the implications of Covid-19, which can potentially have significant health economic effects. For example, the interventions may prolong patients' meaningful activities of daily living and their ability to return to their previous workplaces (conduct their professions). This project will deepen the knowledge about the effects of specialized rehabilitation

Ethical considerations:

The project has been approved by the Swedish Ethical Review Authority. The participants will receive verbal and written information about the study and informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who have undergone Covid-19 and have 80% or less of the lower limit of predicted value in maximal inspiratory pressure (MIP).

Exclusion Criteria:

* Physical och cognitive dysfunction which makes it impossible to carry out measurements and interventions. Already on-going intervention with inspiratory muscle training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Maximal Inspiratory Pressure (MIP) | Measured before and after the intervention period of 8 weeks to detect a change
  Change in MIP measured in cmH20, expressed as percentage of predictive value, with a Respiratory Pressure Meter (Micro RPM)

SECONDARY OUTCOMES:
Change in Maximal Expiratory Pressure (MEP) | Measured before and after the intervention period of 8 weeks to detect a change
  Change in MEP measured in cmH20, expressed as percentage of predictive value, with a Respiratory Pressure Meter (Micro RPM)
Change in Lung function | Measured before and after the intervention period of 8 weeks to detect a change
  Change in Forced Expiratory Volume in one second (FEV1), Forced Vital Capacity (FVC), Peak Expiratory Flow (PEF) and FEV1/FVC measured with spirometry. FEV1 and FVC are measured in liters (l) and PEF in liter/second (l/s). Alla values expressed as percentage of predictive value,
Change in walking distance during 6 minute walk test, expressed as percentage of predictive value, | Measured before and after the intervention period of 8 weeks to detect a change
  Change in walking distance measured in meters during 6 minutes walk test (6MWT)
Change in oxygen saturation during 6 minute walk test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in the lowest oxygen saturation level measured in percentage (%) with pulse oximetry during 6 minute walk test
Change in oxygen desaturation during 6 minute walk test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in drop in percentage points in oxygen saturation during 6 minute walk test. The drop in percentage points is calculated by subtracting the oxygen level at rest before the test with the lowest level during the test.
Change in dyspnea during 6 minute walk test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in perceived dyspnea measured with Borg Category-Ratio scale (Borg CR-10) at the end of 6 minute walk test. Borg CR-10 ranging between 0-10. The higher the score, the higher the dyspnea.
Change in leg fatigue during 6 minute walk test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in perceived leg fatigue measured with Borg CR-10 at the end of 6 minute walk test. Borg CR-10 ranging between 0-10. The higher the score, the higher the leg fatigue.
Change in exertion during 6 minute walk test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in perceived exertion measured with Borg Rating of Perceived Exertion (Borg RPE) at the end of 6 minutes walk test. Borg RPE ranging between 6-20. The higher the score, the higher the exertion.
Change in heart rate during 6 minute walk test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in the highest heart rate measured in beats per minute with pulse oximeter during 6 minute walk test
Change in number of stands in 30 seconds | Measured before and after the intervention period of 8 weeks to detect a change
  Change in number of stands measured during chair stand test after 30 seconds
Change in number of stands in 60 seconds, expressed as percentage of predictive value. | Measured before and after the intervention period of 8 weeks to detect a change
  Change in number of stands measured during chair stand test after 60 seconds
Change in oxygen saturation during chair stand test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in lowest oxygen saturation level measured in percentage (%) with pulse oximetry during chair stand test (60 s)
Change in oxygen desaturation during chair stand test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in drop in percentage points in oxygen saturation during chair stand test. The drop in percentage points is calculated by subtracting the oxygen level at rest before the test with the lowest level during the test.
Change in dyspnea during chair stand test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in perceived dyspnea measured with Borg CR-10 at the end of chair stand test (60 s). Borg CR-10 ranging between 0-10. The higher the score, the higher the dyspnea.
Change in leg fatigue during chair stand test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in perceived leg fatigue measured with Borg CR-10 at the end of chair stand test (60 s). Borg CR-10 ranging between 0-10. The higher the score, the higher the leg fatigue.
Change in exertion during chair stand test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in perceived exertion measured with Borg RPE scale at the end of chair stand test (60 s). Borg RPE scale ranging between 6-20. The higher the score, the higher the exertion.
Change in heart rate during chair stand test | Measured before and after the intervention period of 8 weeks to detect a change
  Change in the highest heart rate measured in beats per minute with pulse oximeter during chair stand test (60 s).
Change in Dyspnea - mMRC (decrease of >= 1) | Measured before and after the intervention period of 8 weeks to detect a change
  Measured with Modified Medical Research Council (mMRC), which is a self-rating tool to measure the degree of disability that breathlessness postures on daily physical activities on a scale from 0 to 4. 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a hill; 2, walks slower than people of same age on the level because of breathlessness; 3, stops for breath when walking at their own pace on the level; and 4, Breathless when washing or getting dressed. A decrease of at least 1 is considerad clinicallty relevant.
Change in Health-related quality of life (EQ5d-index, EQ VAS) | Measured before and after the intervention period of 8 weeks to detect a change
  Measured with EuroQOL 5 dimensions questionnaire (EQ-5D-5L), which is an instrument that evaluates the generic quality of life. EQ-5D includes a descriptive system, which comprises 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A descriptive index-score between 0-1, higher score indicates higher HRQoL. EQ-5D also includes a visual analog scale (VAS), which records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher HRQoL.
Change in Work ability | Measured before and after the intervention period of 8 weeks to detect a change
  Measured with Work Ability Index (WAI), which is a self assessment tool consisting of 7 items. Scores ranging from 7-49. Higher score indicates higher work ability.
Change in Fatigue (FSS-mean score ) | Measured before and after the intervention period of 8 weeks to detect a change
  Measured with Fatigue Severity Scale (FSS), which is a 9-item scale that measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Total score ranging from 9-63. The higher the score, the more severe the fatigue is.
Change in self-reported outcome measure of physical function | Measured before and after the intervention period of 8 weeks to detect a change
  Measured with Patient Specific Functional Scale (PSFS), a questionnaire that can be used to quantify activity limitation and measure functional outcome for patients. Patients are asked to identify three to five important activities they are unable to perform or are having difficulty with because of their problem. In addition to identifying the activities, patients are asked to rate, on a scale ranging from 0-10, the current level of difficulty associated with each activity. The higher the score, the less difficulty to perform the activity.
Change in Voice function | Measured before and after the intervention period of 8 weeks to detect a change
  Measured with a self-assessment form of voice function (SOFT) and a standardized voice recording in a studio. Total score of SOFT ranging between 0-3. Higher score means more difficulties.
Change in Respiratory symptoms | Measured before and after the intervention period of 8 weeks to detect a change
  Respiratory rate visually measured during 60 seconds at rest and self-reported symptoms including chest tightness, impaired deep breathing, and breathing pain
Change in Physical activity (Frändin/Grimby increase of >= 1 level) | Measured before and after the intervention period of 8 weeks to detect a change
  Measured with Frändin/Grimby activity scale, which is a self-assessment scale about current levels of physical activity, ranging from 1 to 6. The higher the score, the higher level of physical activity.
Clinically meaningful improvements in MIP and EQ VAS | Changes between baseline and post-intervention assessment. Eight week intervention period.
  Established minimal clinically important differences (MCIDs) for individuals with PCC were used. MCID for MIP is an increase of at least 22.1%. MCID for EQ VAS is 7.5.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Nygren Bonnier, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No